CLINICAL TRIAL: NCT03726671
Title: Choline Nutritional Status: Development of a Biomarker Panel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 17-1982; 1R01DK115380-01 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-31 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Healthy volunteers will consume meals, provided by the investigator, in two week intervals with 3 different levels of choline (Cho). Participants will receive 100% of the recommended daily intake (RDI) of Cho (550 mg Cho/day); 50% of the RDI of Cho (275mg/day); and 25% of the RDI of Cho (137.5 mg/day). The meal order will be randomly assigned and all participants will receive all diets at some point in the study. There will be a minimum of a two week washout between diet intervals where participants return to their regular diets. Both participants and researchers will be blinded to the diet order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant dietary arm assignment is randomized by a randomization plan created by the study coordinator at www.randomization.com. Each of the 3 hormonal related demographic groups (male, premenopausal females, and postmenopausal females) will have a list of the same order of diets created by the randomizer. Each participant will be assigned upon entry into the study into the next open diet for their group as ordered by the randomizer. No one collecting or processing data will be informed of the choline levels the participant is experiencing in their dietary arms at any given time to attempt to eliminate bias and ensure appropriate data collection. All staff who interact with participants or who are handling samples/data, will not be informed of the code linking dietary choline levels to diet order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25%Cho, 50%Cho, 100%Cho (Experimental): Diets containing 137.5mg (25% Cho diet), 275mg (50% Cho diet), and 550mg (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 25% Cho, 100% Cho, 50% Cho (Experimental): Diets containing 137.5mg (25% Cho diet) , 550mg (100% Cho diet), and 275mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 50% Cho, 25% Cho, 100% Cho (Experimental): Diets containing 275mg (50% Cho diet), 137.5mg (25% Cho diet), and 550mg Cho (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 50% Cho, 100% Cho, 25% Cho (Experimental): Diets containing 275mg (50% Cho diet), 550mg (100% Cho diet), and 137.5mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 100% Cho, 25% Cho, 50% Cho (Experimental): Diets containing 550mg (100% Cho diet), 137.5mg (25% Cho diet), and 275mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 100% Cho, 50% Cho, 25% Cho (Experimental): Diets containing 550mg (100% Cho diet), 275mg (50% Cho diet), and 137.5mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet

INTERVENTIONS:
Other: 25% Cho diet — Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%), Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 137.5mg Choline/day
Other: 50% Cho diet — Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%), Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 275mg Choline/day
Other: 100% Cho diet — Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%), Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 550mg Choline/day

SUMMARY:
People who eat diets low in choline should deplete their choline (Cho) stores, and measurements of Cho pool size using isotope dilution should reflect this depletion. Investigators will identify a biomarker panel that correlates well with measured Cho pool size across the range of different degrees of depletion.The investigators propose that, as body stores of Cho diminish, cells and organs will reach the point when metabolism/function in the cell is altered, and that this will result in a progression of changes in biomarkers that reflect Cho status.

DETAILED DESCRIPTION:
Choline (Cho) is an essential nutrient and most Americans' diets do not achieve the recommended intake. Diets low in Cho are associated with liver and muscle disease and with suboptimal fetal development, while diets too high in choline may be associated with increased risk for heart disease. Cho is a required nutrient and in 1998, an Adequate Intake (AI) and a Tolerable Upper Limit (UL) for Cho was established In 2016, the US Food and Drug Administration (FDA) set a Recommended Daily Intake (RDI) for Cho based on the AIs as part of the new Nutrition Facts label for packaged foods (published in the Federal Register on May 27, 2016; FDA-2012-N-1210-0875, Federal Register Number:2016-11867). The AI/RDI varies by age and gender, but is 550 mg/d in adolescent and adult men and 425 mg/d in adult women (more in pregnant and lactating women) and 400 mg/day for adolescent women.

There is no validated biomarker for choline status (the availability of the various forms of Cho needed to sustain optimal cellular function). Measurement of plasma Cho concentrations is not adequate as plasma choline is homeostatically regulated. Based on extensive preliminary and published data this group identified a panel of potential biomarkers that could be used to assess Cho status, and now the investigators propose to validate this biomarker panel against measures of Cho pool size using isotope dilution. The largest stores of Cho are located in the liver, and mass resonance spectroscopy (MRS) of liver has been used in the past to assess Cho status in humans. This method is not practical for use as a biomarker in clinical or public health practice as it is expensive and the availability of the instrumentation is limited. However, the MRS can be utilized to confirm correlations between the biomarker panel and the isotope dilution method. Liver biopsy is risky and not practical, making measurement of hepatic Cho and Cho metabolites concentrations a poor choice for assessing Cho status.

Perhaps there is a panel of biomarkers that together will more accurately and reliably reflect Cho status. By making measurements in people fed 3 different dietary amounts of Cho for two weeks at a time, and comparing the biomarker measures to body total Cho pool size assessed using isotope dilution (a proxy for the availability of the various forms of Cho), investigators will be able to identify the combination of biomarkers and algorithm for calculating a Cho status score that best predicts total Cho pool size, and therefore predicts choline nutritional status (the availability of the various forms of Cho needed to sustain cellular function). People who eat diets low in choline should deplete their choline (Cho) stores, and measurement of Cho pool size using isotope dilution should reflect this depletion. The investigators will identify a biomarker panel that correlates well with measured Cho pool size across the range of different degrees of depletion. This study tests a method for using stable isotope dilution to measure body choline stores, and then asks how this measure correlates with a panel of biomarkers in plasma and with liver fat measured using Fibroscan®. Using isotope dilution can provide an estimate of the size of the body pool of Cho. The investigators' proposed method is conceptually similar to the method for measuring total body water from a bolus dose of labeled water. Similar methodology was used recently in studies of metabolic flux of Cho in pregnant women. Isotope dilution is a well-established method used to estimate pool size for other nutrients, such as vitamin A. Similar to vitamin A, the major storage pools for Cho are in the liver, and ingested Cho is rapidly absorbed and accumulated by liver. MRS/MRI scans will also be performed to investigate correlation between these "gold standard" measures and the other methods described above.

Participants will consume meals provided in two week dietary intervals with 3 different levels of choline with a 2 week washout periods between those dietary intervals. Participants will receive 100% of the recommended intake (RDI) of Cho (550mg Cho/day); 50% of the RDI of Cho (275mg/day); and 25% of the RDI of Cho (137.5mg/day). The meal order will be randomly assigned and all participants will receive all diets at some point in the study. There will be a minimum of a two week washout between diet intervals. Both participants and researchers will be blinded to the diet order.

Participants will have brief exercise challenges (Biodex) to assess muscle function as an additional predictor of choline status.

Participants enrolled prior to 3/2020 completed MRI/MRS scans. We have determined that Fibroscan provides adequate measurement of liver fat such that we eliminated the added inconvenience to participants of travel to Winston-Salem for MR scanning.

Saliva, stool, and urine samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Weigh 130-177lbs (or if over 177 must have BMI under 28)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 17-70 years
* In good general health as evidenced by medical history, clinical chemistries, physical exam, and BMI≤ 30 or if over 177lbs with a BMI under 28
* Women who are included in the study and are of pregnancy potential will have a urine pregnancy test at the beginning and end of each dietary intervention arm and must be using some form of birth control during the study.

Exclusion Criteria:

* using drugs or medication known to be damaging to liver or muscle at typically prescribed doses or that have the potential to alter Cho metabolism (e.g., methotrexate);
* history of hepatic, renal, or other chronic systemic disease.
* subjects with liver abnormalities (e.g.cysts) as determined by ultrasound
* current smokers
* consume >2 alcoholic beverages/d or >14/wk
* substance abusers or drug addicted
* eating unusual diet that would interfere with the study
* food allergies, (e.g., soy) or any problems with eating all foods on required study diet
* using Cho-containing dietary supplements
* women who are breastfeeding, pregnant, or plan to become pregnant due to potential risk to fetus/child of low choline diet
* performing intense exercise of more than 1 hour a day or other intense muscle building exercise (such as weightlifting beyond low weight repetitions)
* Actively participating in other research study where required to exercise or ingest any food, medicine, or supplement in any manner
* have been screened for this study between August and March and have not provided proof of flu vaccination prior to enrollment

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Zeisel, MD, PhD, Principal Investigator — UNC Chapel Hill - Nutrition Research Institute
Locations (1):
- UNC Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Horita DA, Hwang S, Stegall JM, Friday WB, Kirchner DR, Zeisel SH. Two methods for assessment of choline status in a randomized crossover study with varying dietary choline intake in people: isotope dilution MS of plasma and in vivo single-voxel magnetic resonance spectroscopy of liver. Am J Clin Nutr. 2021 Jun 1;113(6):1670-1678. doi: 10.1093/ajcn/nqaa439. PMID 33668062

RESULTS

PARTICIPANT FLOW:
Groups:
- 25%Cho, 50%Cho, 100%Cho: Diets containing 137.5 mg (25% Cho diet), 275 mg (50% Cho diet), and 550 mg (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
- 25% Cho, 100% Cho, 50% Cho: Diets containing 137.5 mg (25% Cho diet) , 550 mg (100% Cho diet), and 275 mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
- 50% Cho, 25% Cho, 100% Cho: Diets containing 275 mg (50% Cho diet), 137.5 mg (25% Cho diet), and 550 mg Cho (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
- 50% Cho, 100% Cho, 25% Cho: Diets containing 275 mg (50% Cho diet), 550 mg (100% Cho diet), and 137.5 mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
- 100% Cho, 25% Cho, 50% Cho: Diets containing 550 mg (100% Cho diet), 137.5 mg (25% Cho diet), and 275 mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
- 100% Cho, 50% Cho, 25% Cho: Diets containing 550 mg (100% Cho diet), 275 mg (50% Cho diet), and 137.5 mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus
Period: First Intervention (2 Weeks)
Arm/Group | 25%Cho, 50%Cho, 100%Cho | 25% Cho, 100% Cho, 50% Cho | 50% Cho, 25% Cho, 100% Cho | 50% Cho, 100% Cho, 25% Cho | 100% Cho, 25% Cho, 50% Cho | 100% Cho, 50% Cho, 25% Cho
Started | 27 | 14 | 14 | 13 | 24 | 9
Completed | 20 | 12 | 12 | 12 | 19 | 8
Not Completed | 7 | 2 | 2 | 1 | 5 | 1
Period: Washout (>/= 2 Weeks)
Arm/Group | 25%Cho, 50%Cho, 100%Cho | 25% Cho, 100% Cho, 50% Cho | 50% Cho, 25% Cho, 100% Cho | 50% Cho, 100% Cho, 25% Cho | 100% Cho, 25% Cho, 50% Cho | 100% Cho, 50% Cho, 25% Cho
Started | 20 | 12 | 12 | 12 | 19 | 8
Completed | 20 | 12 | 12 | 12 | 19 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | 25%Cho, 50%Cho, 100%Cho | 25% Cho, 100% Cho, 50% Cho | 50% Cho, 25% Cho, 100% Cho | 50% Cho, 100% Cho, 25% Cho | 100% Cho, 25% Cho, 50% Cho | 100% Cho, 50% Cho, 25% Cho
Started | 20 | 12 | 12 | 12 | 19 | 8
Completed | 17 | 12 | 12 | 11 | 18 | 8
Not Completed | 3 | 0 | 0 | 1 | 1 | 0
Period: Washout (>/= 2 Weeks)
Arm/Group | 25%Cho, 50%Cho, 100%Cho | 25% Cho, 100% Cho, 50% Cho | 50% Cho, 25% Cho, 100% Cho | 50% Cho, 100% Cho, 25% Cho | 100% Cho, 25% Cho, 50% Cho | 100% Cho, 50% Cho, 25% Cho
Started | 17 | 12 | 12 | 11 | 18 | 8
Completed | 17 | 12 | 12 | 11 | 17 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | 25%Cho, 50%Cho, 100%Cho | 25% Cho, 100% Cho, 50% Cho | 50% Cho, 25% Cho, 100% Cho | 50% Cho, 100% Cho, 25% Cho | 100% Cho, 25% Cho, 50% Cho | 100% Cho, 50% Cho, 25% Cho
Started | 17 | 12 | 12 | 11 | 17 | 8
Completed | 17 | 11 | 12 | 11 | 17 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Participants: All participants who were randomly assigned to diet sequence containing 137.5 mg (25% Cho diet), 275 mg (50% Cho diet), and 550 mg (100% Cho diet) for two weeks each with 2 weeks of washout between.
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 100
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 85
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101
Menopausal Status [Count of Participants; unit: Participants]
  Pre-Menopausal Females | 50
  Post-Menopausal Females | 21

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Liver Choline Pool Size by Isotope Dilution
Description: The liver choline pool determined by the dilution of the deuterated choline metabolites formed in liver and released to plasma as measured by isotopic enrichment ratio (IER). The IER for a given metabolite is defined as the concentration of a deuterated metabolite divided by the sum of deuterated and non-deuterated metabolite.
Time Frame: 24 hours following administration of choline-d9 on day 12 of respective dietary intervention
Population: Participants who completed at least 2 arms were included in the analysis. Out of 101 randomized, 78 met this criteria. Of the 78, 3 were excluded for noncompliance, leaving 75 participants. Of these 75, 75 completed the 25%, 73 completed the 50% & 75 completed the 100% diets. One participant completing 3 arms was missing 50% isotope dilution data; consequently, outcomes analyzed for 75 participants (25%), 72 participants (50%), & 75 participants (100%).
Measure: Mean (Standard Deviation); unit: isotopic enrichment ratio
Groups:
- 25% Cho: Diet containing 137.5 mg (25% Cho diet) given for two weeks with =/> 2 weeks of washout.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 50% Cho: Diet containing 275 mg Cho (50% Cho diet) given for two weeks with =/> 2 weeks of washout.
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 100% Cho: Diet containing 550 mg Cho (100% Cho diet) given for two weeks each with =/> 2 weeks of washout.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
Arm/Group | 25% Cho | 50% Cho | 100% Cho
Number analyzed (Participants) | 75 | 72 | 75
isotopic enrichment ratio
  Betaine IER | 0.02357 (0.00802) | 0.02403 (0.00882) | 0.02184 (0.00574)
  Choline IER | 0.00023 (0.00511) | 0.00132 (0.00493) | 0.00191 (0.00399)
  Phosphatidylcholine IER | 0.01158 (0.00326) | 0.01130 (0.00324) | 0.01017 (0.00234)
Statistical Analysis 1: Comparison: 25% Cho vs 50% Cho vs 100% Cho; Betaine IER; Test type: Other; p = 0.0247, Repeated measures ANOVA
Statistical Analysis 2: Comparison: 25% Cho vs 50% Cho vs 100% Cho; Choline IER; Test type: Other; p < 0.0001, Repeated measures ANOVA
Statistical Analysis 3: Comparison: 25% Cho vs 50% Cho vs 100% Cho; Phosphatidylcholine IER; Test type: Other; p = 0.0002, Repeated measures ANOVA

2. Primary Outcome: Difference in Choline Deficiency Signature
Description: Plasma choline metabolites (micromolar): choline, dimethylglycine, betaine, phosphatidylcholine, sphingomyelin, trimethylamine-oxide, and homocysteine measured by targeted metabolomic profiling. The signature for choline deficiency is defined by choline <0.793 mmol/L or betaine <34.9 mmol/L. The levels of these metabolites at the end of each intervention will be compared. The association between choline metabolites and choline pool size will be investigated.
Time Frame: At the end of 2 weeks of respective Cho diet
Population: Participants who completed at least 2 arms were included in the analysis. Out of 101 randomized, 78 met this criteria. Of the 78, 3 were excluded for noncompliance, leaving 75 participants. Of these 75, 75 completed the 25%, 73 completed the 50% & 75 completed the 100% diets.
Measure: Number; unit: percentage participants with signature
Arm/Group | 25% Cho | 50% Cho | 100% Cho
Number analyzed (Participants) | 75 | 73 | 75
percentage participants with signature | 57 | 47 | 23
Statistical Analysis 1: Comparison: 25% Cho vs 100% Cho; Test type: Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 7.16, 95% CI 2-sided [3.48 to 14.7]
Statistical Analysis 2: Comparison: 50% Cho vs 100% Cho; Test type: Other; p = 0.01, Fisher Exact; Odds Ratio (OR) = 4.09, 95% CI 2-sided [2.06 to 8.11]
Statistical Analysis 3: Comparison: 25% Cho vs 50% Cho; Test type: Other; p = 0.086, Fisher Exact; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.86 to 3.58]

3. Primary Outcome: Comparison of Choline Pool Size Between Participants With and Without Choline Metabolites Signature During Cho Depletion
Description: The 25% Cho arm was selected because only at that intake level is sufficient depletion achieved. Participants with plasma choline <0.793 mmol/L or betaine <34.9 mmol/L were considered as choline depleted (showing signature), participants with plasma choline >=0.793 mmol/L and betaine >=34.9 mmol/L were considered as not choline depleted (not showing signature). Available choline pool size was determined by the dilution of the deuterated choline metabolites formed in liver and released to plasma as measured by isotopic enrichment ratio (IER). The IER for a given metabolite is defined as the concentration of a deuterated metabolite divided by the sum of deuterated and non-deuterated metabolite.
Time Frame: 24 hours following administration of choline-d9 on day 12 of 25% Cho diet
Population: Participants who completed at least 2 arms were included in the analysis. Out of 101 randomized, 78 met this criteria. Of the 78, 3 were excluded for noncompliance, leaving 75 participants. All 75 participants completed 25% Cho diet. Only data from the 25% Cho diet (choline depleted state) were analyzed.
Measure: Mean (Standard Deviation); unit: isotopic enrichment ratio (uM/uM)
Groups:
- Signature Present During Choline Depletion: A low choline diet (25% Cho) was used to deplete choline pools. The presence of metabolite signature is a sign of choline deficiency.
- Signature Absent During Choline Depletion: A low choline diet (25% Cho) was used to deplete choline pools. Choline deficiency is less likely in the absence of the metabolite signature.
Arm/Group | Signature Present During Choline Depletion | Signature Absent During Choline Depletion
Number analyzed (Participants) | 57 | 18
isotopic enrichment ratio (uM/uM)
  Betaine IER | 0.0234 (0.0087) | 0.0241 (0.0057)
  Choline IER | -0.0005 (0.0049) | 0.0025 (0.0051)
  Phosphatidylcholine IER | 0.0115 (0.0034) | 0.0118 (0.0030)
Statistical Analysis 1: Comparison: Signature Present During Choline Depletion vs Signature Absent During Choline Depletion; Betaine IER; Test type: Other; p = 0.6985, t-test, 2 sided
Statistical Analysis 2: Comparison: Signature Present During Choline Depletion vs Signature Absent During Choline Depletion; Choline IER; Test type: Other; p = 0.0350, t-test, 2 sided
Statistical Analysis 3: Comparison: Signature Present During Choline Depletion vs Signature Absent During Choline Depletion; Phosphatidylcholine IER; Test type: Other; p = 0.6864, t-test, 2 sided

4. Primary Outcome: Ion Abundance (Intensity) of Metabolites as Indicators of the Intake of 25%, 50%, or 100% Choline in the Diet. The Ratio of the Intensity of Metabolite Signals for Each Dietary Group Can be Calculated and Correlated With the Level of Choline in the Diet
Description: Metabolomics was conducted on plasma that was collected from individuals at the end of each 2-week diet period. UHPLC High Resolution Mass Spectrometry was used for differential profiling (PMID: 33415121). Supervised Orthogonal Partial Least Squares Discriminant Analysis was used to determine signals that differentiated the 25% choline dietary group from the 100% choline dietary group. Metabolites that differentiated the 25% and 100% choline dietary groups with variable importance to projection (VIP) >1 and p-value < 0.05 are reported. The signals for these metabolites were matched by retention time, exact mass, and MS/MS to standards run on the same platform. Because this is a differential profiling method (not quantitative), the mean and standard deviation of peak intensities detected on the untargeted platform are reported. Results are reported for the selected metabolites for the 25%, 50%, and 100% choline dietary groups. Ratios can be obtained by division of the intensity data.
Time Frame: At the end of 2 weeks of respective Cho diet
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ion abundance (intensity)
Arm/Group | 25% Cho | 50% Cho | 100% Cho
Number analyzed (Participants) | 75 | 73 | 75
Ion abundance (intensity)
  L-Carnitine | 1228784.33 (306909.00) | 1178435.52 (316249.45) | 1012630.35 (344564.26)
  Propionylcarnitine | 104096.43 (39621.16) | 99820.22 (48710.67) | 80011.86 (38878.77)
  Valerylcarnitine | 94263.17 (36626.32) | 93531.64 (44570.42) | 82582.08 (40040.76)
  Gamma-Muricholic Acid | 4285.05 (5853.57) | 4927.62 (6834.32) | 2519.32 (4817.63)
  Kynurenate | 3200.20 (1562.40) | 3186.66 (1405.28) | 2739.41 (1362.30)
  N-Acetylglycine | 32411.20 (33107.90) | 28421.55 (27012.58) | 26644.26 (26448.88)
  Deoxycholic Acid | 731438.14 (633205.40) | 802858.85 (772625.96) | 600931.15 (509303.07)
  L-Ornithine | 2696.01 (1213.20) | 2684.53 (1338.50) | 2410.86 (1223.70)
  Methylimidazoleacetic Acid | 9875.65 (6304.32) | 10075.93 (5111.30) | 8510.57 (4212.85)
  N6-Acetyl-L-lysine | 24100.04 (7506.44) | 24361.81 (7273.97) | 22522.45 (5552.79)
  DL-2-Aminoadipic Acid | 3088.49 (1065.78) | 3065.37 (1168.13) | 2805.00 (981.61)
Statistical Analysis 1: Comparison: 25% Cho vs 100% Cho; Test type: Equivalence — There are linear combinations of metabolites that differentiate (non-equivalent) the 25% choline diet from the 100% choline diet; p < 0.049, Paired 2-sided t-test; Supervised OPLSDA was used to determine the variable importance to projections of metabolites/signals that differentiated the 25% and 100% choline diet arms

5. Primary Outcome: Comparison of Choline Pool Size Between Participants With Different Genotypes in Phosphatidylethanolamine-N-methyltransferase (PEMT) Single Nucleotide Polymorphism (SNP rs12325817)
Description: DNA was collected and evaluated for the presence of the PEMT SNP rs12325817. Genotypes was measured by real time polymerase chain reaction (RT-PCR). The magnitude of changes in choline pool size as measured by IER at the end of each dietary intervention was compared among subjects with different genotypes in the PEMT SNP. Linear mixed model with repeated measures was performed for each group (healthy males, pre- and postmenopausal females) separately to study the genotype effect and genotype x diet interaction effect on choline pool size.
Time Frame: 24 hours following administration of choline-d9 on day 12 of respective dietary intervention
Population: Participants who completed at least 2 arms were included in the analysis. Out of 101 randomized, 78 met this criteria. Of the 78, 3 were excluded for noncompliance. Of the 75 remaining, one had missing SNP data. One had missing isotope dilution data in 50% Cho. Two subjects did not complete 50% Cho. That brings the sample size down to 74, 71, and 74 for the 25%, 50%, and 100%, respectively. Overall Number of Participants Analyzed includes Pre- and Post-Menopausal Females & Males.
Measure: Mean (Standard Deviation); unit: isotopic enrichment ratio (uM/uM)
Groups:
- 25% Cho, rs12325817, CC: Diet containing 137.5 mg (25% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have CC genotype.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 25% Cho, rs12325817, CG: Diet containing 137.5 mg (25% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have CG genotype.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 25% Cho, rs12325817, GG: Diet containing 137.5 mg (25% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have GG genotype.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 50% Cho, rs12325817, CC: Diet containing 275 mg Cho (50% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have CC genotype.
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 50% Cho, rs12325817, CG: Diet containing 275 mg Cho (50% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have CG genotype.
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 50% Cho, rs12325817, GG: Diet containing 275 mg Cho (50% Cho diet) given for two weeks with =/> 2 weeks of washout. These participants have GG genotype.
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 100% Cho, rs12325817, CC: Diet containing 550 mg Cho (100% Cho diet) given for two weeks each with =/> 2 weeks of washout. These participants have CC genotype.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 100% Cho, rs12325817, CG: Diet containing 550 mg Cho (100% Cho diet) given for two weeks each with =/> 2 weeks of washout. These participants have CG genotype.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 100% Cho, rs12325817, GG: Diet containing 550 mg Cho (100% Cho diet) given for two weeks each with =/> 2 weeks of washout. These participants have GG genotype.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
Arm/Group | 25% Cho, rs12325817, CC | 25% Cho, rs12325817, CG | 25% Cho, rs12325817, GG | 50% Cho, rs12325817, CC | 50% Cho, rs12325817, CG | 50% Cho, rs12325817, GG | 100% Cho, rs12325817, CC | 100% Cho, rs12325817, CG | 100% Cho, rs12325817, GG
Number analyzed (Participants) | 17 | 34 | 23 | 16 | 34 | 21 | 17 | 34 | 23
isotopic enrichment ratio (uM/uM)
  Pre-Menopausal Females: Betaine IER: number analyzed (Participants) | 11 | 17 | 10 | 10 | 17 | 10 | 11 | 17 | 10
  Pre-Menopausal Females: Betaine IER | 0.0259 (0.0101) | 0.0201 (0.01) | 0.0261 (0.0064) | 0.0244 (0.0073) | 0.0224 (0.0059) | 0.0262 (0.0073) | 0.0243 (0.0072) | 0.0213 (0.0046) | 0.0247 (0.0039)
  Pre-Menopausal Females: Choline IER: number analyzed (Participants) | 11 | 17 | 10 | 10 | 17 | 10 | 11 | 17 | 10
  Pre-Menopausal Females: Choline IER | -0.0018 (0.0051) | -0.0018 (0.0063) | -0.0011 (0.0028) | -0.0004 (0.0051) | 0.0004 (0.0054) | -0.0007 (0.0036) | 0.0004 (0.0044) | 0.0008 (0.0042) | 0.0001 (0.0039)
  Pre-Menopausal Females: Phosphatidylcholine IER: number analyzed (Participants) | 11 | 17 | 10 | 10 | 17 | 10 | 11 | 17 | 10
  Pre-Menopausal Females: Phosphatidylcholine IER | 0.0113 (0.003) | 0.011 (0.0044) | 0.011 (0.0024) | 0.011 (0.0027) | 0.011 (0.0032) | 0.0115 (0.0033) | 0.0107 (0.0024) | 0.0105 (0.0025) | 0.01 (0.0017)
  Post-Menopausal Females: Betaine IER: number analyzed (Participants) | 3 | 6 | 5 | 3 | 6 | 4 | 3 | 6 | 5
  Post-Menopausal Females: Betaine IER | 0.0212 (0.007) | 0.02 (0.0033) | 0.0265 (0.0124) | 0.0136 (0.0126) | 0.0212 (0.0026) | 0.028 (0.0127) | 0.0232 (0.0037) | 0.0175 (0.0026) | 0.02 (0.0086)
  Post-Menopausal Females: Choline IER: number analyzed (Participants) | 3 | 6 | 5 | 3 | 6 | 4 | 3 | 6 | 5
  Post-Menopausal Females: Choline IER | 0.0014 (0.0048) | -0.0001 (0.0039) | 0.0017 (0.005) | 0.0006 (0.0084) | 0.0007 (0.0042) | 0.0044 (0.0045) | 0.0047 (0.0022) | 0.0019 (0.0027) | 0.0026 (0.0035)
  Post-Menopausal Females: Phosphatidylcholine IER: number analyzed (Participants) | 3 | 6 | 5 | 3 | 6 | 4 | 3 | 6 | 5
  Post-Menopausal Females: Phosphatidylcholine IER | 0.0095 (0.0021) | 0.009 (0.0014) | 0.0127 (0.0043) | 0.0071 (0.0049) | 0.01 (0.001) | 0.0121 (0.0041) | 0.0096 (0.0016) | 0.0086 (0.0011) | 0.0096 (0.0023)
  Males: Betaine IER: number analyzed (Participants) | 3 | 11 | 8 | 3 | 11 | 7 | 3 | 11 | 8
  Males: Betaine IER | 0.0264 (0.0059) | 0.025 (0.0053) | 0.024 (0.0045) | 0.0419 (0.0264) | 0.0241 (0.0045) | 0.0222 (0.0021) | 0.0247 (0.0053) | 0.0201 (0.0077) | 0.0213 (0.0036)
  Males: Choline IER: number analyzed (Participants) | 3 | 11 | 8 | 3 | 11 | 7 | 3 | 11 | 8
  Males: Choline IER | 0.0043 (0.0026) | 0.0029 (0.0034) | 0.003 (0.0061) | 0.0097 (0.0022) | 0.0028 (0.0026) | 0.0029 (0.0045) | 0.0061 (0.0005) | 0.0029 (0.0038) | 0.0041 (0.0042)
  Males: Phosphatidylcholine IER: number analyzed (Participants) | 3 | 11 | 8 | 3 | 11 | 7 | 3 | 11 | 8
  Males: Phosphatidylcholine IER | 0.0131 (0.0002) | 0.0135 (0.0021) | 0.013 (0.0027) | 0.0184 (0.0034) | 0.0111 (0.0019) | 0.0123 (0.0016) | 0.0127 (0.0007) | 0.0094 (0.0035) | 0.0112 (0.0012)
Statistical Analysis 1: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Betaine IER in Pre-Menopausal Females; Test type: Other; p = 0.9567, Mixed Models Analysis; The model evaluates effects from SNP, diet and SNP x diet interaction. Due to crossover design, period and sequence effects were adjusted in the model
Statistical Analysis 2: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Betaine IER in Post-Menopausal Females; Test type: Other; p = 0.0899, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Betaine IER in Males; Test type: Other; p = 0.9003, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Choline IER in Pre-Menopausal Females; Test type: Other; p = 0.9932, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Choline IER in Post-Menopausal Females; Test type: Other; p = 0.3984, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Choline IER in Males; Test type: Other; p = 0.3080, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Phosphatidylcholine IER in Pre-Menopausal Females; Test type: Other; p = 0.7603, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Phosphatidylcholine IER in Post-Menopausal Females; Test type: Other; p = 0.2995, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; Diet x SNP interaction effect on Phosphatidylcholine IER in Males; Test type: Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Betaine IER in Pre-Menopausal Females; Test type: Other; p = 0.1303, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Betaine IER in Post-Menopausal Females; Test type: Other; p = 0.0015, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Betaine IER in Males; Test type: Other; p = 0.4185, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Choline IER in Pre-Menopausal Females; Test type: Other; p = 0.3464, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 14: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Choline IER in Post-Menopausal Females; Test type: Other; p = 0.0019, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 15: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Choline IER in Males; Test type: Other; p = 0.2091, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 16: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Phosphatidylcholine IER in Pre-Menopausal Females; Test type: Other; p = 0.8141, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 17: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Phosphatidylcholine IER in Post-Menopausal Females; Test type: Other; p = 0.0187, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 18: Comparison: 25% Cho, rs12325817, CC vs 25% Cho, rs12325817, CG vs 25% Cho, rs12325817, GG vs 50% Cho, rs12325817, CC vs 50% Cho, rs12325817, CG vs 50% Cho, rs12325817, GG vs 100% Cho, rs12325817, CC vs 100% Cho, rs12325817, CG vs 100% Cho, rs12325817, GG; SNP effect on Phosphatidylcholine IER in Males; Test type: Other; p = 0.0107, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]

6. Primary Outcome: Change in Liver Fat Content Based on CAP Values
Description: Controlled attenuation parameter (CAP) as measured by Fibroscan is an ultrasound-based technique to measure liver fat. This method will be used with other biomarkers to indicate functional signs of choline status.
Time Frame: Day 1 and Day 15 of respective Cho diet
Population: Participants who completed at least 2 arms were included in the analysis. Out of 101 randomized, 78 met this criteria. Of the 78, 3 were excluded for noncompliance, leaving 75 participants. Of these 75, 75 completed the 25%, 73 completed the 50% & 75 completed the 100% diets. Fibroscan data were missing for 2 participants in the 25% Cho arm and 2 in the 50% arm.
Measure: Mean (Standard Deviation); unit: dB/m
Arm/Group | 25% Cho | 50% Cho | 100% Cho
Number analyzed (Participants) | 73 | 71 | 75
dB/m | 0.0208 (0.1513) | 0.6958 (0.2144) | 0.0135 (0.1482)
Statistical Analysis 1: Comparison: 25% Cho vs 50% Cho vs 100% Cho; Test type: Other; p = 0.0842, Mixed Models Analysis
Statistical Analysis 2: Comparison: 25% Cho vs 50% Cho; Test type: Other; p = 0.0819, Wilcoxon (Mann-Whitney); Non-parametric method was used due to data deviation from normality
Statistical Analysis 3: Comparison: 25% Cho vs 100% Cho; Test type: Other; p = 0.9015, t-test, 2 sided
Statistical Analysis 4: Comparison: 50% Cho vs 100% Cho; Test type: Other; p = 0.1191, Wilcoxon (Mann-Whitney); Non-parametric method was used due to data deviation from normality

7. Secondary Outcome: Validation of Isotope Dilution Method to Assess Choline Pool Size by Magnetic Resonance Spectroscopy (MRS)
Description: MRS is a direct measurement of liver choline content. Changes in liver choline by MRS should correlate with changes in liver choline inferred by calculation of isotope enrichment ratio (IER) of plasma metabolites. Pearson correlation coefficient used to study the correlation between data generated from the two types of measurements.
Time Frame: At the end of 2 weeks of respective Cho diet
Population: MRS was run on only an initial 40 participants due to limited funding. Due to extensive variation, MRS data were not usable for 8 participants in the 25%, 10 participants in the 50%, and 8 participants in the 100% Cho arms.
Measure: Mean (Standard Deviation); unit: mM
Groups:
- 25%Cho: Diet containing 137.5 mg (25% Cho diet) given for two weeks with =/> 2 weeks of washout.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride (trimethyl-d9, 9%) as a bolus.
- 100% Cho: Diets containing 550mg Cho (100% Cho diet) will be given for two weeks with =/> 2 weeks of washout.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride-(trimethyl-d9, 9% as a bolus
Arm/Group | 25%Cho | 50% Cho | 100% Cho
Number analyzed (Participants) | 32 | 30 | 32
mM | 8.4 (4.1) | 7.8 (4.5) | 11.2 (7.2)
Statistical Analysis 1: Comparison: 25%Cho vs 100% Cho; Liver choline concentration vs. betaine IER; Test type: Other; p = 0.2351, Pearson's Correlation Coefficient
Statistical Analysis 2: Comparison: 25%Cho vs 100% Cho; Liver choline concentration vs. Phosphatidylcholine IER; Test type: Other; p = 0.4501, Pearson's Correlation Coefficient
Statistical Analysis 3: Comparison: 25%Cho vs 100% Cho; Liver choline concentration vs. Choline IER; Test type: Other; p = 0.4136, Pearson's Correlation Coefficient
Statistical Analysis 4: Comparison: 50% Cho vs 100% Cho; Liver choline concentration vs. Betaine IER; Test type: Other; p = 0.9463, Pearson's Correlation Coefficient
Statistical Analysis 5: Comparison: 50% Cho vs 100% Cho; Liver choline concentration vs. Phosphatidylcholine IER; Test type: Other; p = 0.0675, Pearson's Correlation Coefficient
Statistical Analysis 6: Comparison: 50% Cho vs 100% Cho; Liver choline concentration vs. Choline IER; Test type: Other; p = 0.2863, Pearson's Correlation Coefficient
Statistical Analysis 7: Comparison: 25%Cho vs 50% Cho; Liver choline concentration vs. Betaine IER; Test type: Other; p = 0.5552, Pearson's Correlation Coefficient
Statistical Analysis 8: Comparison: 25%Cho vs 50% Cho; Liver choline concentration vs. Phosphatidylcholine IER; Test type: Other; p = 0.4209, Pearson's Correlation Coefficient
Statistical Analysis 9: Comparison: 25%Cho vs 50% Cho; Liver choline concentration vs. Choline IER; Test type: Other; p = 0.6647, Pearson's Correlation Coefficient

8. Other Pre Specified Outcome: SNPs That Create Inefficiencies in Choline Metabolism Associated With Change in Choline Pool Size and Choline Biomarkers
Description: Exploratory analysis of >2 million SNPs measured on a custom Illumina Expanded Multi-Ethnic genotyping array (Mega-Ex). The same analysis described for Outcome 4 will be applied for Outcome 7. Benjamini-Hochberg method for False Discovery Rate (FDR) correction will be used for multiple testing correction.
Time Frame: At baseline visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of informed consent throughout the duration of a participant's involvement in the study, a combined total of approximately 10 weeks
Groups:
- 25% Cho: Diets containing 137.5 mg (25% Cho diet) will be given for two weeks.
  25% Cho diet: Subjects will consume meals containing 25% of recommended intake of Choline for 2 weeks.
- 50% Cho: Diets containing 275 mg Cho (50% Cho diet) will be given for two weeks.
  50% Cho diet: Subjects will consume meals containing 50% of recommended intake of Choline for 2 weeks.
- 100% Cho: Diets containing 550 mg Cho (100% Cho diet) will be given for two weeks.
  100% Cho diet: Subjects will consume meals containing 100% of recommended intake of Choline for 2 weeks.
Arm/Group | 25% Cho | 50% Cho | 100% Cho
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/84 | 0/86
Other Adverse Events (participants affected / at risk) | 0/91 | 0/84 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03726671/Prot_SAP_000.pdf